CLINICAL TRIAL: NCT07228325
Title: A Comparison of PK and PD Responses Following Single and Repeat Administration of Epinephrine Nasal FMXIN002 4.0 mg and EpiPen 0.3 mg, in Healthy Adults With Allergic Rhinitis
Brief Title: Comparative PK/PD of FMXIN002 and EpiPen, in Healthy Adults With Allergic Rhinitis
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nasus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP-007-Epinephrine
Record Dates: First submitted 2025-11-06; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Anaphylaxis; Allergy
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FMXIN002 Repeated doses in the same nostril (Experimental): Repeated doses of epinephrine nasal powder spray, in the same nostril, 10 minutes apart.
  Interventions: Drug: FMXIN002 single dose; Drug: Epinephrine autoinjector single dose; Drug: FMXIN002 single dose + NAC; Drug: Epinephrine autoinjector double dose; Drug: FMXIN002 double dose; Drug: FMXIN002 double dose + NAC
- FMXIN002 Repeated doses in the opposite nostril (Experimental): Repeated doses of epinephrine nasal powder spray, in both nostrils, 10 minutes apart.
  Interventions: Drug: FMXIN002 single dose; Drug: Epinephrine autoinjector single dose; Drug: FMXIN002 single dose + NAC; Drug: Epinephrine autoinjector double dose; Drug: FMXIN002 double dose; Drug: FMXIN002 double dose + NAC

INTERVENTIONS:
Drug: FMXIN002 single dose — Single dose of FMXIN002 epinephrine microspheres powder for nasal application, 4.0 mg, at normal conditions.
  Other Names: NS002
Drug: Epinephrine autoinjector single dose — Epinephrine IM autoinjector 0.3mg
  Other Names: EpiPen
Drug: FMXIN002 single dose + NAC — Single dose of FMXIN002 epinephrine microspheres powder for nasal application, 4.0 mg, after Nasal Allergenic Challenge (NAC)
  Other Names: NS002
Drug: Epinephrine autoinjector double dose — Repeated doses of Epinephrine IM autoinjector 0.3mg, 10 minutes apart
  Other Names: EpiPen
Drug: FMXIN002 double dose — Double doses of FMXIN002 epinephrine microspheres powder for nasal application, 4.0 mg, at normal conditions, 10 minutes apart.
  Other Names: NS002
Drug: FMXIN002 double dose + NAC — Double doses of FMXIN002 epinephrine microspheres powder for nasal application, 4.0 mg, after Nasal Allergenic Challenge, 10 minutes apart.
  Other Names: NS002

SUMMARY:
The study will evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) responses of FMXIN002, an intranasal epinephrine powder, compared with the EpiPen® intramuscular autoinjector, after single and double doses, in healthy adults with a history of allergic rhinitis.

DETAILED DESCRIPTION:
Fifty participants will receive single and repeat doses of both treatments under normal and nasal congestion conditions induced by nasal allergen challenge. The study will also assess the effect of repeat nasal dosing in the same versus opposite nostrils. PK parameters and hemodynamic responses will be measured, and safety and tolerability will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, male and female participants, from 18 to 55 years of age.
2. Documented positive skin allergy test at screening.
3. History of hay fever, seasonal allergies, or allergic rhinitis during the last year.
4. BMI ≥18 and < =30 kg/m2.
5. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:

     o Physically capable of becoming pregnant, must be willing to use acceptable effective methods of contraception.
   * Non-childbearing potential:

     * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or
     * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause and a FSH value consistent with being postmenopausal).
6. Able to tolerate venipuncture.
7. Be informed of the nature of the study and give written consent prior to any study procedure.
8. Willing and able to remain in the clinic for the entire duration of the confinement period.
9. Have good intravenous access on both arms and hands. -

Exclusion Criteria:

* History of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study results.
* Have clinically significant findings at screening.
* Females who:

  * Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to the first drug administration;
  * Have discontinued or changed the use of oral or patch hormonal contraceptives within one (1) month prior to the first drug administration;
  * Are pregnant (serum β-hCG consistent with pregnancy); or
  * Are breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Epinephrine level in plasma over time | -60 to 240 minutes post administration
  Measurements in 14 timepoints
Tmax | -60 to 240 minutes post administration
  Time to maximum epinephrine level in plasma
T100pg/ml | -60 to 240 minutes post administration
  Time to reach epinephrine level of 100pg/ml in plasma
Cmax | -60 to 240 minutes post administration
  Maximum epinephrine level in plasma
AUC | 0 to 240 minutes post administration
  Total exposure to epinephrine
Blood pressure | -60 to 120 minutes post administration
  Pharmacodynamic response to epinephrine
Heart rate | -60 to 120 minutes post administration
  Pharmacodynamic response to epinephrine
Respiratory rate | -60 to 120 minutes post administration
  Pharmacodynamic response to epinephrine

SECONDARY OUTCOMES:
Safety and tolerability | Day -29 to day 50
  Adverse events rate at each treatment, and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Freedman, MD, FRCPC, Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Research Inc, Mississauga, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will share documents as required by the future scientific journal of choice.